CLINICAL TRIAL: NCT01145066
Title: Modulation of Biomarkers and Gene Expression by Botanical Oil Supplementation in Diabetic and Metabolic Syndrome Subjects.
Brief Title: Botanical Oil Supplementation in Diabetic and Metabolic Syndrome Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00007488; P50 AT 0027820 (Other Grant/Funding Number: NCCAM)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Metabolic Syndrome x
Keywords: diabetes; metabolic syndrome; inflammation; botanical oils
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Inflammation | interventions — Fish Oils; lanpol 5; Corn Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- borage and echium oil combination (Experimental): borage/echium oil combination containing 0.85g/day SDA and 1.7 g/day GLA
  Interventions: Drug: borage/echium oil combination
- fish oil (Active Comparator): Croda 18:12 fish oil
  Interventions: Dietary Supplement: fish oil
- corn oil (Placebo Comparator)
  Interventions: Dietary Supplement: corn oil

INTERVENTIONS:
Drug: borage/echium oil combination — borage/echium oil combination containing 0.85g/day SDA and 1.7g/day GLA
  Other Names: Croda echium oil SR06379; Croda borage oil, Crossential GLA TG40
  Arms: borage and echium oil combination
Dietary Supplement: fish oil — 1.6g/day EPA and 1.08g/day DHA
  Other Names: Croda 18:12 fish oil
  Arms: fish oil
Dietary Supplement: corn oil — contains 4.5 g/day linoleic acid
  Other Names: Croda superrefined corn NF
  Arms: corn oil

SUMMARY:
This study will compare how well a combination of borage and echium oils will reduce inflammation compared to fish oils and placebo oil in subjects that are diabetic or have metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* adults, aged 21 years or more with either diabetes or metabolic syndrome. metabolic syndrome defined by NCEP/ATPIII criteria; must have 3 out of 5 of the following risk factors: 1.central obesity, men-greater than or equal to 40 inches, women-greater than or equal to 35 inches; 2.fasting blood TG greater than or equal to 150mg/dl or be taking TG lowering medications; 3. blood HDL cholesterol, men less than 40 mg/dl, women less than 50 mg/dl; 4. blood pressure greater than or equal to 130/85 or on HTN medication 5. fasting glucose greater than or equal to 100 mg/dl.
* participants on statins or glucose lowering drugs if dosages are stable for 3 months

Exclusion criteria

* children/young adults less than 21 years of age
* currently using anti-inflammatory drugs including NSAIDS, oral/IV steroids or injection antiinflammatory drugs(for RA), aspirin greater than 100mg/day
* taking leukotriene receptor antagonists ( montelukast), tylenol or nasal/inhaled steroids OK.
* currently using niacin, fibrates or fish oil
* blood pressure greater than 170/100
* HB1Ac greater than 10%
* TG greater than 500 mg/dl
* myocardial infarction/vascular surgery/stroke within the past year
* any stage II,III,IV heart failure
* prior cholecystectomy
* end stage renal disease
* BMI less than 23 or greater than 45
* pregnancy
* alcohol use greater than 14 drinks per week
* current self reported tobacco or illicit drug use
* intolerance or allergy to fish oil
* participants taking insulin on QD or BID doses, stable for 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Floyd(Ski) H Chilton, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Lee TC, Ivester P, Hester AG, Sergeant S, Case LD, Morgan T, Kouba EO, Chilton FH. The impact of polyunsaturated fatty acid-based dietary supplements on disease biomarkers in a metabolic syndrome/diabetes population. Lipids Health Dis. 2014 Dec 16;13:196. doi: 10.1186/1476-511X-13-196. PMID 25515553

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 participants signed consent, only 71 were randomized to an arm/group
Period: Overall Study
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Started | 26 | 20 | 25
Completed | 22 | 16 | 21
Not Completed | 4 | 4 | 4
Not completed — To resume NSAIDs | 2 | 2 | 1
Not completed — Non-related surgery | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — To start new med | 1 | 0 | 0
Not completed — problems swallowing capsule | 1 | 0 | 0
Not completed — Abdominal discomfort | 0 | 1 | 0
Not completed — Low platelet count | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil | Total
Number analyzed (Participants) | 22 | 16 | 21 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (7.8) | 56.2 (8.7) | 59.9 (9.8) | 57.96 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 15 | 35
  Male | 12 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Fasting Insulin
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
μIU/mL | 15.4 (2.0) | 19.1 (4.5) | 20.2 (3.2)

2. Primary Outcome: Fasting Insulin
Description: Fasting insulin data at 4 and 8 weeks was averaged.
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
μIU/mL | 17.7 (2.6) | 24.6 (6.8) | 20.6 (3.3)

3. Primary Outcome: hsCRP
Description: Changes in high sensitive C-reactive protein (hsCRP) were assessed.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/L | 3.03 (.85) | 6.08 (3.19) | 2.36 (.57)

4. Primary Outcome: hsCRP
Description: Changes in high sensitive C-reactive protein (hsCRP) were assessed and data at 4 and 8 weeks was averaged..
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/L | 3.06 (.86) | 3.59 (1.03) | 3.72 (1.00)

5. Primary Outcome: Leptin
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
ng/mL | 33.3 (6.2) | 45.1 (11.0) | 53.5 (6.8)

6. Primary Outcome: Leptin
Description: Data at 4 and 8 weeks was averaged.
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
ng/mL | 33.9 (7.4) | 40.6 (7.2) | 44.2 (5.3)

7. Secondary Outcome: Serum Fatty Acids
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage of total fatty acids
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
percentage of total fatty acids
  Cl4:0 | .69 (.08) | .72 (.07) | .70 (.07)
  C14:1 | 0 (0) | 0 (0) | 0 (0)
  C15:0 | .13 (.02) | .16 (.02) | .15 (.02)
  C15:1 | 0 (0) | 0 (0) | 0 (0)
  C16:0 | 20.64 (.41) | 21.65 (.47) | 21.19 (.40)
  C16:1 n-7 | 1.58 (.08) | 1.92 (.24) | 1.68 (.13)
  C17:1 | .10 (.02) | .13 (.03) | .08 (.02)
  C18:0 | 7.23 (.14) | 7.00 (.25) | 7.47 (.09)
  C18:1 | .12 (.07) | .17 (.06) | .21 (.06)
  C18:1 n-9 | 19.6 (.44) | 21.92 (.98) | 20.63 (.96)
  C18:1 n-11 | 1.5 (.07) | 1.84 (.06) | 1.60 (.06)
  C18:2 n-6 [LA] | 32.67 (.98) | 29.71 (1.28) | 31.99 (1.26)
  C18:3 n-6 [GLA] | .59 (.04) | .55 (.05) | .53 (.03)
  C18:3 n-3 [ALA] | .80 (.05) | .77 (.09) | .73 (.06)
  C18:4 n-3 [SDA] | .01 (.01) | .01 (.01) | .03 (.02)
  C20:0 | 0 (0) | 0 (0) | .01 (.01)
  C20:1 n-9 | .04 (.01) | .10 (.02) | .08 (.02)
  C20:2 n-6 | .32 (.01) | .33 (.02) | .30 (.02)
  C20:3 n-6 [DGLA] | 1.51 (.08) | 1.43 (.09) | 1.68 (.08)
  C20:4 n-6 [AA] | 9.12 (.40) | 8.68 (.40) | 8.17 (.56)
  C20:5 n-3 [EPA] | .573 (.05) | .56 (.07) | .48 (.04)
  C22:0 | 0 (0) | 0 (0) | 0 (0)
  C22:1 n-9 | .15 (.06) | 0 (0) | .05 (.04)
  C22:2 n-6 | 0 (0) | 0 (0) | 0 (0)
  C22:5 n-3 [DPA] | .55 (.02) | .59 (.03) | .54 (.03)
  C24:0 | .02 (.02) | 0 (0) | .02 (.02)
  C22:6 n-3 [DHA] | 1.63 (.10) | 1.73 (.016) | 1.71 (.12)
  C24:1 n-9 | .01 (.01) | .04 (.02) | .03 (.02)

8. Secondary Outcome: Serum Fatty Acids
Description: Data at 4 and 8 weeks was averaged.
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: percentage of total fatty acids
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
percentage of total fatty acids
  Cl4:0 | .66 (.04) | .62 (.06) | .66 (.05)
  C14:1 | 0 (0) | 0 (0) | 0 (0)
  C15:0 | .14 (.02) | .14 (.02) | .14 (.02)
  C15:1 | 0 (0) | 0 (0) | 0 (0)
  C16:0 | 20.49 (.37) | 20.76 (.39) | 20.75 (.37)
  C16:1 n-7 | 1.39 (.08) | 1.55 (.14) | 1.57 (.13)
  C17:1 | .05 (.02) | .06 (.02) | .04 (.02)
  C18:0 | 7.55 (.16) | 7.39 (.27) | 7.62 (.12)
  C18:1 | .13 (.05) | .25 (.06) | .25 (.05)
  C18:1 n-9 | 19.60 (.44) | 20.24 (.52) | 20.30 (.61)
  C18:1 n-11 | 1.44 (.05) | 1.56 (.06) | 1.51 (.06)
  C18:2 n-6 [LA] | 30.97 (.80) | 29.94 (1.14) | 33.11 (.93)
  C18:3 n-6 [GLA] | 1.2 (.08) | .45 (.05) | .52 (.03)
  C18:3 n-3 [ALA] | 1.05 (.05) | .83 (.06) | .71 (.05)
  C18:4 n-3 [SDA] | .08 (.01) | .02 (.01) | .01 (0)
  C20:0 | 0 (0) | 0 (0) | .01 (0)
  C20:1 n-9 | .04 (.01) | .03 (.01) | .05 (.01)
  C20:2 n-6 | .24 (.01) | .23 (.18) | .31 (.01)
  C20:3 n-6 [DGLA] | 1.97 (.09) | 1.45 (.07) | 1.61 (.05)
  C20:4 n-6 [AA] | 9.16 (.34) | 7.31 (.36) | 8.11 (.46)
  C20:5 n-3 [EPA] | .89 (.08) | 2.79 (.18) | .46 (.05)
  C22:0 | 0 (0) | 0 (0) | 0 (0)
  C22:1 n-9 | .15 (.06) | .19 (.11) | .11 (.04)
  C22:2 n-6 | 0 (0) | 0 (0) | 0 (0)
  C22:5 n-3 [DPA] | .55 (.02) | .89 (.03) | .51 (.03)
  C24:0 | .01 (.01) | .01 (.01) | .02 (.01)
  C22:6 n-3 [DHA] | 1.63 (.10) | 3.58 (.11) | 1.60 (.11)
  C24:1 n-9 | 0 (0) | 0 (0) | .01 (.01)

9. Secondary Outcome: Pro and Anti-inflammatory Cytokines
Time Frame: baseline
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Pro and Anti-inflammatory Cytokines
Time Frame: 4 weeks and 8 weeks combined
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Fasting Glucose
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/dL | 125.9 (7.3) | 133.5 (16.7) | 130.0 (9.8)

12. Secondary Outcome: Fasting Glucose
Description: Data at 4 and 8 weeks was averaged.
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/dL | 125.9 (1.09) | 128.7 (11.1) | 130.7 (11.2)

13. Secondary Outcome: Hemoglobin Levels
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/dL | 6.81 (.30) | 7.42 (.33) | 7.15 (.34)

14. Secondary Outcome: Hemoglobin Levels
Description: Data at 4 and 8 weeks was averaged.
Time Frame: 4 weeks and 8 weeks combined
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 22 | 16 | 21
mg/dL | 6.90 (.27) | 7.20 (.32) | 7.07 (.35)

15. Secondary Outcome: Adipose Derived Cytokines
Time Frame: 4 weeks
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: PBMC Gene Expression
Time Frame: baseline
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: PBMC Gene Expression
Time Frame: 4 weeks
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: SNPs in DNA of Selected Genes
Time Frame: baseline
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: SNPs in DNA of Selected Genes
Time Frame: 4 weeks
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: PBMC Leukotriene Stimulation
Time Frame: baseline
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: PBMC Leukotriene Stimulation
Time Frame: 4 weeks
Population: No data collected
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Borage and Echium Oil Combination | Fish Oil | Corn Oil
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/20 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/20 | 0/25
Other Adverse Events (participants affected / at risk) | 4/26 | 5/20 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Borage and Echium Oil Combination (N=26) | Fish Oil (N=20) | Corn Oil (N=25)
Sick/virus (Immune system disorders) | 3 | 3 | 3
GI Upset (Gastrointestinal disorders) | 0 | 0 | 2 — Bloating/constipation
GI Upset (Gastrointestinal disorders) | 0 | 1 | 0 — burping/diarrhea/loose stools
Headache (Nervous system disorders) | 1 | 0 | 0
Weak (Metabolism and nutrition disorders) | 0 | 1 | 1 — blood sugar varied 1 day or more

LIMITATIONS AND CAVEATS:
The diet study was short at only 8 weeks of oil supplementation, it did not control background PUFA consumption by the subjects throught their normal diets, and the population contained subjects at various stages of T2D.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes